CLINICAL TRIAL: NCT06170736
Title: Radiofrequency Haemorrhoidal Thermoablation Versus Doppler-guided Haemorrhoidal Artery Ligation With Mucopexy in the Treatment of Haemorrhoidal Disease: a Multicenter Randomized Non-inferiority Trial
Brief Title: Radiofrequency Ablation vs Doppler-guided Haemorrhoidal Artery Ligation in the Treatment of Haemorrhoidal Disease
Acronym: RADIOLIGA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Departemental Vendee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHD22_0066
Record Dates: First submitted 2023-12-06; First posted 2023-12-14 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Haemorrhoids; Internal Haemorrhoids; Grade II/III Haemorrhoids
Keywords: Haemorrhoids; Radiofrequency; Doppler-guided haemorrhoidal artery ligation
MeSH Terms: conditions — Hemorrhoids | interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Doppler-Guided Haemorrhoidal Artery Ligation (Active Comparator): Patients will be treated by DGHAL procedure.
  Interventions: Procedure: Doppler-Guided Haemorrhoidal Artery Ligation
- Radiofrequency Ablation (Experimental): Patients will be treated by radiofrequency ablation.
  Interventions: Procedure: Radiofrequency ablation

INTERVENTIONS:
Procedure: Doppler-Guided Haemorrhoidal Artery Ligation — The principle consists of locating the signal emitted by the haemorrhoidal arteries using a Doppler probe. Once identified, the arteries are ligated in order to remove the arterial vascularization of the haemorrhoidal bundles. The treatment of the prolapse is reinforced by a folding of the mucosa of the lower rectum, called mucopexy.
  Arms: Doppler-Guided Haemorrhoidal Artery Ligation
Procedure: Radiofrequency ablation — The principle consists of inserting a metal probe under the mucosa of the anus, in contact with the haemorrhoidal bundles to be treated. A source of radiofrequency is then delivered through this probe in contact with the haemorrhoidal veins which will be sclerosed. The procedure is repeated for each haemorrhoidal bundle to be treated.
  Arms: Radiofrequency Ablation

SUMMARY:
Surgical treatment of grade II/III internal haemorrhoidal disease is indicated in the case of medical and/or instrumental treatment failure. Minimal invasive alternatives to haemorrhoidectomy have been introduced in the last decades to treat grade II/III haemorrhoids. Doppler-Guided haemorrhoidal artery ligation (DGHAL) represents a good therapeutic option in this condition with good short and mid-term outcomes but postoperative recurrence rates up to 35% at 5 years.

Recently, a technique of radiofrequency ablation (RFA) has been introduced with promising outcomes. A recent systematic review reported a significant improvement of preoperative symptoms and a recurrence rate < 5%.

To date, there is no study comparing DGHAL to RFA in the treatment of grade II/III haemorrhoids.

The aim of this study is to demonstrate the non-inferiority in terms of failure rate of haemorrhoidal radiofrequency ablation compared to Doppler-guided haemorrhoidal artery ligation, associated with mucopexy, in the treatment of grade II and III haemorrhoidal disease

ELIGIBILITY:
Inclusion Criteria:

* Major patient,
* With symptomatic Grade II or III haemorrhoidal disease,
* Requiring surgical management,
* Patient able to understand the protocol and having given written informed consent to participate in the study,
* Patient affiliated to the social security system or entitled to it.

Exclusion Criteria:

* Hemostasis disorders
* Active external haemorrhoidal disease (thrombosis)
* History of surgical procedure for treatment of haemorrhoids (instrumental treatment is not a contra-indication)
* Associated proctological pathology (anal fissure, chronic suppuration, external rectal prolapse)
* History of colorectal cancer
* History of inflammatory bowel disease
* History of rectal resection
* Patient participating in another interventional clinical research protocol involving a drug or clinical investigation of a medical device
* Patient who is pregnant, breastfeeding or able to procreate without effective contraception* at the time of inclusion
* Patient under guardianship, curators or deprived of liberty.
* Patient under court protection.

  * oral contraceptive (pill), monthly vaginal ring, weekly transdermal patch, subcutaneous implant, intrauterine devices (IUD), or sterilisation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2024-02-21 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2028-09-15 (Estimated)

PRIMARY OUTCOMES:
Failure rate at one year post-operatively | one year post-operatively
  The evaluation of failure rate will be based on the calculation of the HDSS score grouping the different symptoms (pain, discomfort, bleeding, soiling and prolapse). Failure rate will be defined by a score greater than or equal to the preoperative score or by a reoperation (surgical or instrumental) for relapse of the symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Marc-Henri JEAN, Dr, Principal Investigator — Centre Hospitalier Departemental Vendée
Locations (16):
- France (16):
  - Centre Hospitalier Universitaire, Amiens
  - Centre Hospitalier Universitaire, Angers
  - Maison de Santé Bagatelle, Bordeaux
  - Centre Hospitalier Privé, Brest
  - Centre Hospitalier Départemental de Vendée, La Roche-sur-Yon
  - Hôpital de la Louvière, Lille
  - Clinique de la Sauvegarde, Lyon
  - Centre Hospitalier Universitaire, Nantes
  - Clinique Jules Verne, Nantes
  - Hôpital Saint Joseph, Paris
  - Institut Mutualiste Montsouris, Paris
  - Centre Hospitalier Interrégional, Poissy
  - Centre Hospitalier Universitaire, Rennes
  - Cabinet de Proctologie, Saint-Herblain
  - hôpital d'Instruction des Armées, Saint-Mandé
  - Clinique de l'Estuaire, Saint-Nazaire

IPD SHARING:
Plan to Share IPD: No